CLINICAL TRIAL: NCT03215303
Title: Effects of Continuous Positive Airway Pressure (CPAP) on Exercise Capacity of Children and Adolescents With Severe Therapy-resistant Asthma
Brief Title: Effects of CPAP in Severe Therapy-resistant Asthma
Acronym: CPAP-STRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marcio Vinicius Fagundes Donadio, Professor, Pontificia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CPAP
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: Asthma; Continuous positive airway pressure; Oxygen consumption
MeSH Terms: conditions — Asthma | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized, through a sealed envelope, to initially compose the intervention group or the control group. The sequential order of randomization will be kept confidential with a single investigator, so that the other professionals involved and responsible for data collection will be blinded throughout the study period. Individuals who initially composed the intervention group will then perform, in a second moment, the procedures of the control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization process will be kept confidential with a single investigator, not involved in data collection or recruitment, so that all other investigators involved will be blinded to the experimental groups throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Positive Airway Pressure (CPAP) (Experimental): Participants in the intervention group will use CPAP device, for a period of 40 minutes, with the following parameters: PEEP of 10cmH2O and FiO2 0.21.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- CONTROL (Placebo Comparator): Participants in the control group will use CPAP device, for a period of 40 minutes, with the following parameters: PEEP of 1cmH2O and FiO2 0.21.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — In the first moment, CPAP will be installed, and the researcher will hold a mask in the position in which it is coherent, explaining the method to the patient and allowing their gradual adaptation. Patients will adapt for a few minutes to make sure the mask is consistent with the specifications, so that the patient is comfortable. Participants in the intervention group will start with a PEEP of 1cmH2O that will increase by 2 cmH2O until a PEEP of 10 cmH2O is reached. Therefore, participants in the intervention group will remain with CPAP, PEEP of 10cmH2O, FiO2 0.21, for a period of 40 minutes.

SUMMARY:
The purpose of this study is to verify the effects of continuous positive airway pressure (CPAP) on exercise capacity of children and adolescents with severe therapy-resistant asthma (STRA). A randomized, controlled, crossover clinical trial will be conducted. We expect the use of CPAP to increase exercise capacity in children and adolescents with STRA.

DETAILED DESCRIPTION:
This project aims to verify the effects of continuous positive airway pressure (CPAP) on exercise capacity of children and adolescents with severe asthma therapy-resistant (STRA). A randomized, controlled, crossover clinical trial will be conducted. Children and adolescents between 6 and 18 years old, with a diagnosis of STRA, will be included in the study. Patients wil be recruited in the São Lucas Hospital (HSL) Asthma Outpatient Clinic of the Pontifical Catholic University of Rio Grande do Sul. Patients who accept to participate in the study will perform a medical consultation according to routine outpatient asthma clinic, anthropometric evaluation and pulmonary function tests. Afterwards, they will be randomized into control and intervention groups. Participants in the intervention group will use noninvasive ventilation (NIV) in CPAP mode with 10cmH2O of positive end-expiratory pressure (PEEP), fraction of inspired oxygen (FiO2) of 0.21, for a period of 40 minutes. Participants in the control group will use NIV (CPAP), with a minimum PEEP of 1cmH20 and a FiO2 of 0.21 also for 40 minutes. Afterwards, patients from both groups will perform a maximum cardiopulmonary exercise test (CPET). A sample size of 18 individuals to be included in the study was estimated. The variables studied will be maximal oxygen consumption and the anaerobic threshold (that measures exercise capacity), distance and time (to measure exercise tolerance), peripheral oxygen saturation, peak expiratory flow and the sensation of dyspnea at the end of the CPET.

ELIGIBILITY:
Inclusion Criteria:

- Individuals with a clinical diagnosis of severe therapy-resistant asthma (STRA), of both sexes, aged between 6 and 18 years, who are under regular follow-up in the asthma outpatient clinic at São Lucas Hospital, PUCRS.

The criteria for the classification of STRA is based on the Global Initiative for Asthma (GINA) guidelines:

* Asthma requiring treatment in steps 4-5 of GINA (≥800 mg/day of budesonide or equivalent, associated with long-acting ß2-adrenergic agonist (LABA);
* Use of continuous oral corticoid or omalizumab, presenting uncontrolled disease;
* Uncontrolled disease characterized by: 1) persistent symptoms or asthma control test (ACT) <20 (> 3 months); 2) acute exacerbations (with intensive care unit admission, at least 2 hospitalizations, or 2 courses of oral corticoid over the last 12 months); Or 3) non-reversible obstruction of pulmonary function, even after corticoid use.

Exclusion Criteria:

- Subjects with cognitive/motor limitations or other chronic diseases (neurological diseases, cardiac anomalies, congenital or immunodeficiencies), which may compromise the evaluation of asthma, as well as the procedures proposed by the present study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Immediately after intervention
  Exercise capacity will be assessed by the VO2max, evaluated during a cardiopulmonary exercise test. Gas capture measurement will be performed by an ergospirometric system using a VO2000 (Medical Graphics Corporation, St. Paul, Minnesota-USA) gas analyzer, which provides information on ventilatory variables every 20s.

SECONDARY OUTCOMES:
Exercise tolerance | Immediately after intervention
  Exercise tolerance will be assessed by measuring distance in the cardiopulmonary exercise test.
Exercise duration | Immediately after intervention
  Exercise tolerance will be assessed by measuring time in the cardiopulmonary exercise test.
Peripheral oxygen saturation | Immediately after intervention
  Peripheral oxygen saturation will be evaluated at rest, every 60s and at the end of the CPET using a portable pulse oximeter (Nonin®, Minneapolis, USA).
Peak expiratory flow | Immediately after intervention
  Peak expiratory flow will be assessed using a peak flow meter immediately after CPET.
Subjective feeling of dyspnea | Immediately after intervention
  Subjective feeling of dyspnea will be evaluated using the Modified Borg Scale, which uses a graduation from 0 to 10, at the end of the CPET.

CONTACTS AND LOCATIONS:
Overall Officials: Marcio VF Donadio, PHD, Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul
Locations (1):
- Pontifífia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bateman ED, Hurd SS, Barnes PJ, Bousquet J, Drazen JM, FitzGerald JM, Gibson P, Ohta K, O'Byrne P, Pedersen SE, Pizzichini E, Sullivan SD, Wenzel SE, Zar HJ. Global strategy for asthma management and prevention: GINA executive summary. Eur Respir J. 2008 Jan;31(1):143-78. doi: 10.1183/09031936.00138707. PMID 18166595
- [Background] Worldwide variation in prevalence of symptoms of asthma, allergic rhinoconjunctivitis, and atopic eczema: ISAAC. The International Study of Asthma and Allergies in Childhood (ISAAC) Steering Committee. Lancet. 1998 Apr 25;351(9111):1225-32. PMID 9643741
- [Background] McDonald VM, Vertigan AE, Gibson PG. How to set up a severe asthma service. Respirology. 2011 Aug;16(6):900-11. doi: 10.1111/j.1440-1843.2011.02012.x. PMID 21692918
- [Background] Jang AS, Lee JH, Park SW, Shin MY, Kim DJ, Park CS. Severe airway hyperresponsiveness in school-aged boys with a high body mass index. Korean J Intern Med. 2006 Mar;21(1):10-4. doi: 10.3904/kjim.2006.21.1.10. PMID 16646558
- [Background] O'Donnell DE, Sanii R, Giesbrecht G, Younes M. Effect of continuous positive airway pressure on respiratory sensation in patients with chronic obstructive pulmonary disease during submaximal exercise. Am Rev Respir Dis. 1988 Nov;138(5):1185-91. doi: 10.1164/ajrccm/138.5.1185. PMID 3059891
- [Background] Wang CH, Lin HC, Huang TJ, Yang CT, Yu CT, Kuo HP. Differential effects of nasal continuous positive airway pressure on reversible or fixed upper and lower airway obstruction. Eur Respir J. 1996 May;9(5):952-9. doi: 10.1183/09031936.96.09050952. PMID 8793457
- [Background] Busk M, Busk N, Puntenney P, Hutchins J, Yu Z, Gunst SJ, Tepper RS. Use of continuous positive airway pressure reduces airway reactivity in adults with asthma. Eur Respir J. 2013 Feb;41(2):317-22. doi: 10.1183/09031936.00059712. Epub 2012 Jul 26. PMID 22835615
- [Background] Pianosi PT, Davis HS. Determinants of physical fitness in children with asthma. Pediatrics. 2004 Mar;113(3 Pt 1):e225-9. doi: 10.1542/peds.113.3.e225. PMID 14993581
- [Background] Ferrazza AM, Martolini D, Valli G, Palange P. Cardiopulmonary exercise testing in the functional and prognostic evaluation of patients with pulmonary diseases. Respiration. 2009;77(1):3-17. doi: 10.1159/000186694. Epub 2009 Jan 14. PMID 19145106
- [Background] Hallstrand TS, Bates PW, Schoene RB. Aerobic conditioning in mild asthma decreases the hyperpnea of exercise and improves exercise and ventilatory capacity. Chest. 2000 Nov;118(5):1460-9. doi: 10.1378/chest.118.5.1460. PMID 11083702
- [Background] Chatkin M, Menezes AM, Albernaz E, Victora CG, Barros FC. [Asthmatic children's risk factors for emergency room visits, Brazil]. Rev Saude Publica. 2000 Oct;34(5):491-8. doi: 10.1590/s0034-89102000000500009. Portuguese. PMID 11105113
- [Background] Schuh C, Fritscher LG, Chapman KR, Fritscher CC. The prevalence of asthma and atopy in schoolchildren from Porto Alegre, Brazil, has plateaued. Respir Med. 2015 Mar;109(3):308-11. doi: 10.1016/j.rmed.2015.01.014. Epub 2015 Jan 31. PMID 25683031
- [Background] Barbosa e Silva O, Saraiva LC, Sobral Filho DC. Treadmill stress test in children and adolescents: higher tolerance on exertion with ramp protocol. Arq Bras Cardiol. 2007 Dec;89(6):391-7. English, Portuguese. PMID 18317622
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Santuz P, Baraldi E, Filippone M, Zacchello F. Exercise performance in children with asthma: is it different from that of healthy controls? Eur Respir J. 1997 Jun;10(6):1254-60. doi: 10.1183/09031936.97.10061254. PMID 9192925